CLINICAL TRIAL: NCT04855227
Title: ASPIRE: A proSpective Evaluation of PaIn After Non-complex ventRal hErnia Repair
Brief Title: A Prospective Evaluation of Pain After Non-complex Ventral Hernia Repair
Acronym: ASPIRE
Status: Terminated | Type: Observational
Why Stopped: Slow rate of enrollment . Additionally it was observed during the course of the trial that changes to the standard of care pain management protocols at some of the institutions, which are not aligned with the study protocol requirements
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ASPIRE
Record Dates: First submitted 2021-03-30; First posted 2021-04-22 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic ventral hernia repair: These subjects will undergo a laparoscopic primary umbilical or incisional hernia repair.
- Robotic-assisted ventral hernia repair: These subjects will undergo a robotic-assisted primary umbilical or incisional hernia repair.
  Interventions: Procedure: robotic-assisted ventral hernia repair

INTERVENTIONS:
Procedure: robotic-assisted ventral hernia repair — Laparoscopic ventral hernia repair With the subject under general anesthesia, several small incisions are made in the abdomen. Ports are placed, the abdomen is insufflated, and laparoscopic instruments as well as a laparoscope are inserted to complete the repair. The retrorectus space is developed for mesh placement to repair the defect. The repair technique will be per the surgeon's standard of care.
  Robotic-assisted ventral hernia repair With the patient under general anesthesia, several small incisions are made in the abdomen. Ports are placed, the abdomen is insufflated, and the da Vinci Robotic Surgical System (Intuitive) is docked to the subject and used to complete the procedure. The retrorectus space is developed for mesh placement to repair the defect. The repair technique will be per the surgeon's standard of care.
  Other Names: laparoscopic ventral hernia repair
  Groups: Robotic-assisted ventral hernia repair

SUMMARY:
The study aims to evaluate outcomes relating to pain and QOL after robotic-assisted or laparoscopic non-complex ventral hernia repair.

DETAILED DESCRIPTION:
This is a prospective, observational, study across robotic-assisted and laparoscopic primary (non-recurrent) umbilical and incisional hernia repair. The study aims to evaluate pain and QOL outcomes through 30 days. During the post-operative period through 30 days, pain medication intake, subject reported pain and quality of life and incidence of intra-operative and post-operative adverse events related to the ventral hernia repair will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 80 years of age.
2. Subject is a candidate for an elective primary (non-recurrent) ventral hernia repair.
3. Ventral hernia repair that will require mesh placement

Exclusion Criteria:

1. Subject is contraindicated for general anesthesia or surgery.
2. Subject with a ventral hernia that will require retromuscular mesh placement or employ a technique, including (but not limited to) external oblique release, Rives- Stoppa, eTEP Rives-Stoppa, transversus abdominis release, other component separation techniques (i.e. anterior component separation) or eTEP transversus abdominis release.
3. Subject has a recurrent hernia.
4. Subject who will have an emergent hernia repair.
5. Subject with a history of chronic pain and/or taking daily pain medications for >6 weeks.
6. Subject with a history of substance abuse (excluding marijuana) and/or current (within 30 days) narcotic use.
7. Current marijuana use that the subject is unwilling to discontinue within the 14 days prior to surgery.
8. Subject with a history of MRSA infection.
9. Subject with HbA1c level > 8.5%.
10. Use of Exparel during the surgical procedure.
11. Subject who will undergo a concomitant hernia repair or any other concomitant procedure.
12. Current nicotine use (including vaping) within the past 30 days.
13. Subject has a known bleeding or clotting disorder.
14. Pregnant or suspected pregnancy.
15. Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent.
16. Subject belonging to other vulnerable population, e.g, prisoner or ward of the state.
17. Subject is currently participating in another interventional or investigational research study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who will undergo an elective non-complex ventral hernia repair procedure and who meet all eligibility criteria will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Change in pain score assessed by the PROMIS 3a from baseline to 14 days | 14 days
  Change in patient reported pain scores assessed by the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey, with a scale from 1-5; 1 meaning no pain and 5 meaning severe pain.
Change in narcotic usage from 1 day post-procedure to 14 days post-procedure | 14 days
  Narcotic usage after the ventral hernia repair as determined through use of a patient reported pain medication log.
Change in pain score assessed by the NRS from baseline to 14 days | 14 days
  Change in patient reported pain scores assessed by the Numeric Rating Scale (NRS) from 1-10, where 0 indicates no pain and 10 indicates the worst pain imaginable.

SECONDARY OUTCOMES:
Change in narcotic usage from 1 day post-procedure to 30 days post-procedure | 30 days
  Narcotic usage after the ventral hernia repair as determined through use of a patient reported pain medication log.
Change in OTC pain medication usage from 1 day post-procedure to 30 days post-procedure | 30 days
  Over the counter (OTC) pain medication usage after the ventral hernia repair as determined through use of a patient reported pain medication log.
Need for refill prescription pain medication usage from 1 day post-procedure to 30 days post-procedure | 30 days
  Need for refill narcotic prescription pain medication usage
Change in Quality of Life assessment: EQ-5D-3L (EQ) from baseline to 14 days | 14 days
  Quality of life assessment using the EQ-5D-3L (EQ) assessment tool, with scores on individual questions ranging from no problems to extreme problems, with a scale of health ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine)
Change in Quality of Life assessment: EuraHS-QOL from baseline to 30 days | 30 days
  Quality of life using the EuraHS-QOL assessment tool, with scores on questions relating to pain, restrictions of movement, and cosmetic discomfort; with a scale ranging from 0 (no pain/no restriction/very beautiful) to 10 (worst pain/completely restricted/extremely ugly).
Length of hospital stay (LOS) | Procedure start time to discharge from the hospital (check out time), up to an approximate of one week
  How long the patient was admitted to the hospital
Incidence of intraoperative adverse events related to the ventral hernia repair | Intraoperative
  Intraoperative adverse events related to the ventral hernia repair
Incidence of postoperative adverse events related to the ventral hernia repair through 30 days post-procedure | 30 days
  Post-operative adverse events related to the ventral hernia repair

CONTACTS AND LOCATIONS:
Locations (1):
- Desert Surgical Specialists, Phoenix, Arizona, United States